CLINICAL TRIAL: NCT03293251
Title: Trabeculectomy With MMC and I Stent in Uveitic Glaucoma and POAG : Outcomes and Prognostic Factors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Collaborators: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Maha omar mahmoud said, principle investigator, Assiut University
Other Study IDs: 1111
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Outcomes of Trabeculectomy With MMC
MeSH Terms: interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- uveitic/ POAG: Outcomes, success rates, complications of trabeculectomy with MMC in Uveitic glaucoma
  Interventions: Procedure: Trabeculectomy with MMC
- POAG: Outcomes, success rates, complications of trabeculectomy with MMC and I stent in this groups
  Interventions: Procedure: Trabeculectomy with MMC

INTERVENTIONS:
Procedure: Trabeculectomy with MMC — glaucoma surgeries
  Other Names: I-STENT

SUMMARY:
1. determine whether cataract surgery has a major effect on outcomes of trabeculectomy with MMC or not.
2. Success rates of trabeculectomy with MMC in Queen Elizabeth hospital.
3. recurrence rate of uveitis after glaucoma surgery

DETAILED DESCRIPTION:
1. determine different success rates of trabeculectomy with MMC undergone in QE hospital, UK.
2. determine different complications and effect of cataract surgery on the outcome of glaucoma surgery

ELIGIBILITY:
Inclusion Criteria:

* Fesh trabeculectomy surgeries

Exclusion Criteria:

* recurrent surgeries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cohort of patient documented on the database system of Queen Elizabeth hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-29 (Estimated); Study Completion 2018-12-29 (Estimated)

PRIMARY OUTCOMES:
Success rates | 5 year period
  IOP less 21 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kamel Soliman, professor, Study Director — Assiut University
Locations (1):
- Maha Said, Egypt, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided yet